CLINICAL TRIAL: NCT01624272
Title: The Effectiveness of Pranayama Breathing Exercises vs. Threshold Inspiratory Muscle Trainer to Improve Respiratory Muscle Function in an Institutionalized Frail Elderly Population
Brief Title: Respiratory Muscle Training in Institutionalized Elderly Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Maria dels Angels Cebria i Iranzo, PT, PhD, Assistant Professor Rehabilitation Sciences, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: H1325072291220
Record Dates: First submitted 2012-06-13; First posted 2012-06-20 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Muscle Weakness; Syndrome; Institutionalization; Other Diagnoses, Comorbidities, and Complications
Keywords: Physical Therapy; Respiratory Muscle Training; Elderly
MeSH Terms: conditions — Muscle Weakness; Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): Usual care
- Threshold Inspiratory Muscle Training (Experimental): Inspiratory muscle training regime
  Interventions: Device: Threshold® Inspiratory Muscle Trainer (Respironics® Health Scan Inc. Cedar Grove, NJ, USA).
- Controlled breathing exercises (Experimental): Yoga Pranayama breathing exercises
  Interventions: Other: Yoga Pranayama breathing exercises

INTERVENTIONS:
Device: Threshold® Inspiratory Muscle Trainer (Respironics® Health Scan Inc. Cedar Grove, NJ, USA). — Interval-based program consisting of seven cycles of 2-minutes work and 1-minute rest. The sessions took place 5 times per week over a six-week period for a total of 30 sessions. All participants were familiarized with the breathing exercises over a two-day familiarization period at the beginning of the protocol.
  Other Names: Threshold IMT
  Arms: Threshold Inspiratory Muscle Training
Other: Yoga Pranayama breathing exercises — Interval-based program. The sessions took place 5 times per week over a six-week period for a total of 30 sessions. All participants were familiarized with the breathing exercises over a two-day familiarization period at the beginning of the protocol.
  Other Names: Pranayama
  Arms: Controlled breathing exercises

SUMMARY:
The global loss of muscle mass and strength associated with aging is a cause of functional impairment and disability, particularly in the frail elderly. Respiratory function can be severely compromised if there is a decrease of respiratory (RM) strength complicated by the presence of comorbidities and physical immobility.

Previous studies have shown that the specific RM training is an effective method to increase RM strength, both in healthy people and patients. In this case, specific RM training may be regarded as a beneficial alternative to improve RM function, and thus prevent physical and clinical deterioration in this population.

The hypothesis is that specific RM training would improve RM strength and endurance in the experimental groups vs. control who do not participate in RM training.

Institutionalized elderly people with an inability to walk were randomly allocated to a control group, a Threshold group or a Pranayama group. Both experimental groups performed a supervised RM training, five days a week for six consecutive weeks. The maximum inspiratory and expiratory pressures (MIP and MEP) and the maximum voluntary ventilation (MVV) were assessed at four time points in each of three groups.

DETAILED DESCRIPTION:
Studies have shown that general aerobic exercise training is accompanied by significant respiratory physiological benefits, including gains in RM strength and endurance (Larson, et al., 1999; Sheel, 2002; Watsford, et al., 2005; Lacasse et al., 2006). This benefit appears to be greater when general exercise conditioning is combined with specific RM training (Weiner, et al., 1992; Wanke, et al., 1994; Larson, et al., 1999; Hill y Eastwood, 2005; O'Brien, et al., 2008). However, many frail elderly are not able to perform general aerobic exercise, related or not to ADL, as it is mentioned above (e.g., institutionalized elderly with comorbidities, functional impairment and RM weakness). In this case, specific RM training may be used as a beneficial alternative to maintain or improve RM function (Watsford and Murphy, 2008), and thus prevent deterioration in this functionally impaired elderly.

The most commonly used techniques of specific RM training are: a) isocapnic hyperpnoea (Leith and Bradley, 1976; Belman and Mittman, 1980), b) respiratory resistive loading (Pardy, et al., 1981; Sonne and Davis, 1982; Belman, et al., 1986), and c) respiratory threshold loading (Clanton, et al., 1985; Chen, et al., 1985; Martyn, et al., 1987; Larson, et al., 1988). Apart from these three well-known techniques, other less studied types of exercise such as the controlled breathing exercises of Yoga, Pranayama, may also be added to this list (Kulpati, et al., 1982; Manocha, et al., 2002; Donesky-Cueco, et al., 2009).

ELIGIBILITY:
Inclusion Criteria:

* clinically stable residents, institutionalized at least 1 year;
* Barthel Index less than 95 points;
* inability to independently walk more than 10 meters or inability to effectively use a wheelchair;
* Mini-Mental Status Examination score of at least 20 points (i.e., subjects without moderate or severe cognitive deterioration).

Exclusion Criteria:

* significant chronic cardiorespiratory diagnoses (e.g. moderate-severe COPD);
* an acute cardiorespiratory episode during the last 2 months prior to the study;
* neurological, muscular, or neuromuscular problems interfering with the capacity to engage in the tests and training protocols;
* active smokers or former smokers who had stopped smoking less than 5 years ago;
* a terminal disease.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Maximum Inspiratory Pressure (MIP) at 7 weeks | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 7).
  MIP is probably the most frequently reported noninvasive estimates of inspiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal inspiration. The manoeuvre is generally performed at Residual Volume (RV). Reference: Am J Respir Crit Care Med. 2002;166:531-535.
Change from baseline in Maximum Expiratory Pressure (MEP) at 7 weeks | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 7).
  MEP is probably the most frequently reported noninvasive estimates of expiratory muscle strength. Ever since Black and Hyatt (1969) reported this technique it has been widely used in patients, healthy control subjects across all ages, and athletes. Pressure is recorded at the mouth during a quasi-static short (few seconds) maximal expiration. The manoeuvre is generally performed at Total Lung Capacity (TLC). Reference: Am J Respir Crit Care Med. 2002;166:531-535.

SECONDARY OUTCOMES:
Change from baseline in Maximum Voluntary Ventilation at 7 weeks | The groups were assessed at baseline (time zero) and at the end of the training protocol (week 7).
  This ventilatory test is a non-invasive technique and is a measure of both inspiratory and expiratory muscle endurance. The MVV is the largest volume that can be breathed in and out of the lungs during a 12 -15 second interval with maximal voluntary effort. Reference: Am J Respir Crit Care Med. 2002;166:562-564.

CONTACTS AND LOCATIONS:
Overall Officials: M. Àngels Cebrià i Iranzo, PT, PhD, Principal Investigator — University of Valencia; David A Arnall, PT, PhD, Study Chair — East Tennessee State University; Celedonia Igual Camacho, PT, PhD, Study Chair — University of Valencia; José M Tomás, PhD, Study Chair — University of Valencia
Locations (3):
- Spain (3):
  - Residencia de la Tercera Edad "San Luis", Moncada, Valencia
  - Residencia de la Tercera Edad "El Amparo", Quart de Poblet, Valencia
  - Ballesol- Centros residenciales 3ª edad, Valencia, Valencia

REFERENCES:
- [Result] Cebria I Iranzo MD, Arnall DA, Igual Camacho C, Tomas JM, Melendez JC. Physiotherapy intervention for preventing the respiratory muscle deterioration in institutionalized older women with functional impairment. Arch Bronconeumol. 2013 Jan;49(1):1-9. doi: 10.1016/j.arbres.2012.07.007. Epub 2012 Sep 19. English, Spanish. PMID 22999331
- [Result] Cebria i Iranzo Md, Arnall DA, Igual Camacho C, Tomas JM. Effects of inspiratory muscle training and yoga breathing exercises on respiratory muscle function in institutionalized frail older adults: a randomized controlled trial. J Geriatr Phys Ther. 2014 Apr-Jun;37(2):65-75. doi: 10.1519/JPT.0b013e31829938bb. PMID 23835773
- [Result] Cebria I Iranzo MD, Tortosa-Chulia MA, Igual-Camacho C, Sancho P, Galiana L, Tomas JM. [Cost-consequence analysis of respiratory preventive intervention among institutionalized older people: randomized controlled trial]. Rev Esp Geriatr Gerontol. 2014 Sep-Oct;49(5):203-9. doi: 10.1016/j.regg.2013.11.002. Epub 2014 Jan 11. Spanish. PMID 24417971